CLINICAL TRIAL: NCT06284850
Title: Red Blood Cell 2,3-biphosphoglycerate Levels in Patients Treated With Empagliflozin. A Prospective Cohort Study.
Brief Title: Empagliflozin and Red Blood Cell 2,3-biphosphoglycerate Levels
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Christina Trakatelli, Assistant Professor Of Internal Medicine, Aristotle University Of Thessaloniki
Other Study IDs: Christina Trakatelli
Record Dates: First submitted 2024-01-10; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hematocrit Change; Cardiovascular Prevention; Empagliflozin; SGLT2-Inhibitors; Tissue Oxygenation
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- treatment with empagliflozin 10mg od: empagliflozin 10mg OD
  Interventions: Drug: Empagliflozin10Mg Tab

INTERVENTIONS:
Drug: Empagliflozin10Mg Tab — TB JARDIANCE 10MG
  Other Names: JARDIANCE 10MG

SUMMARY:
The aim of this study is to investigate the hypothesis that treatment with empagliflozin may have an impact on red blood cell 2,3-biphosphoglycerate levels affecting tissue oxygen supply and thus mediating part of the cardio- and reno- protective effect of SGLT-2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

Patients>18 year-old and at least one of the following

* Type 2 Diabetes Mellitus and HbA1c: 6.5-9.0% or HbA1c <6.5% and history of Coronary Artery Disease or Stroke not treated with GLP-1RA
* Heart Failure defined as Ejection Fraction<40% or NT-proBNP>300pg/ml or Atrial fibrillation and NT-proBNP>900pg/ml
* Chronic Kidney Disease defined as eGFR<60ml/min/1.73m2 (CKPD- EPI) or/and UACR>200mg/g Initiating treatment with empagliflozin 10mg once daily as add on treatment

Exclusion Criteria:

* Patients already treated with an SGLT-2 inhibitor
* Patients with Hb<11gr/dl or>16gr/dl
* Patients with history of inherited or acquired hemoglobin disease
* Patients with history of hemolytic anemia
* Patients with history of hematologic malignancy or myelodysplastic syndrome or myeloproliferative syndrome
* Patients treated within the last 6 months for anemia due to iron, B12 or folate deficiency
* Patients with history of major hemorrhage or major operation leading to RBC transfusion within the last 3 months.
* Patients planning major operation or revascularization procedure within the 12 following weeks
* Patients treated with erythropoietin
* Patients with Chronic Kidney Disease and GFR<30ml/min/1.73m2
* Pregnancy
* Women of childbearing age not receiving appropriate contraception measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients>18 year-old and at least one of the following
  * Type 2 Diabetes Mellitus and HbA1c: 6.5-9.0% or HbA1c <6.5% and history of Coronary Artery Disease or Stroke not treated with GLP-1RA
  * Heart Failure defined as Ejection Fraction<40% or NT-proBNP>300pg/ml or Atrial fibrillation and NT-proBNP>900pg/ml
  * Chronic Kidney Disease defined as eGFR<60ml/min/1.73m2 (CKPD- EPI) or/and UACR>200mg/g Initiating treatment with empagliflozin 10mg once daily as add on treatment
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mean change in red blood cell 2,3-biphosphoglycerate levels (μmol/ml) | 12 weeks
  Mean change in red blood cell 2,3-biphosphoglycerate levels (μmol/ml)

SECONDARY OUTCOMES:
Mean change in Hct (%) | 12 weeks
  Mean change in Hct(%)
Hb (mg/dl) | 12 weeks
  Mean change in Hb (mg/dl)
RBC (x1000000/μl) | 12 weeks
  Mean change in RBC (x1000000/μl)
MCV (fl), | 12 weeks
  Mean change in MCV (fl)
HbA1c (%, mmol/mol), | 12 weeks
  Mean change inHbA1c (%, mmol/mol)
erythropoietin (mU/ml) | 12 weeks
  Mean change in erythropoietin (mU/ml)
eGFR (ml/min/1.73m2), | 12 weeks
  Mean change in eGFR (ml/min/1.73m2),
Urine Albumin to Creatinine Ratio (mg/g) | 12 weeks
  Mean change in Urine Albumin to Creatinine Ratio (mg/g)

CONTACTS AND LOCATIONS:
Overall Officials: KONSTANTINOS KITSIOS, MD,MSc,PhD, Principal Investigator — Aristotle University of Thessaloniki 3d Department of Internal Medicine, Papageorgiou General Hospital, Thessaloniki, Greece
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided
concerns about personal data safety